CLINICAL TRIAL: NCT00025038
Title: Phase II Window Evaluation of the Farnesyl Transferase Inhibitor (R115777) Followed by 13-CIS Retinoic Acid, Cytosine Arabinoside and Fludarabine Plus Hematopoietic Stem Cell Transplantation in Children With Juvenile Myelomonocytic Leukemia
Brief Title: Combination Chemotherapy Followed By Donor Bone Marrow or Umbilical Cord Blood Transplant in Treating Children With Newly Diagnosed Juvenile Myelomonocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01861; AAML0122; U10CA098543 (NIH); CDR0000068788 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2001-10-11; First posted 2003-01-27 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-01

CONDITIONS: Juvenile Myelomonocytic Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Juvenile | interventions — tipifarnib; Isotretinoin; fludarabine phosphate; Cytarabine; Radiotherapy; Radiation; Cyclophosphamide; Antilymphocyte Serum; thymoglobulin; Transplantation; Cord Blood Stem Cell Transplantation

ARMS (1):
- Treatment (tipifarnib, bone marrow/umbilical cord transplant) (Experimental): See detailed description.
  Interventions: Drug: tipifarnib; Drug: isotretinoin; Drug: fludarabine phosphate; Drug: cytarabine; Radiation: radiation therapy; Drug: cyclophosphamide; Biological: anti-thymocyte globulin; Procedure: allogeneic bone marrow transplantation; Procedure: double-unit umbilical cord blood transplantation; Procedure: umbilical cord blood transplantation; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: tipifarnib — Given orally
  Other Names: R115777; Zarnestra
Drug: isotretinoin — Given orally
  Other Names: 13-CRA; Amnesteem; Cistane; Claravis; Sotret
Drug: fludarabine phosphate — Given IV
  Other Names: 2-F-ara-AMP; Beneflur; Fludara
Drug: cytarabine — Given IV
  Other Names: ARA-C; arabinofuranosylcytosine; arabinosylcytosine; Cytosar-U; cytosine arabinoside
Radiation: radiation therapy — Undergo total body irradiation
  Other Names: irradiation; radiotherapy; therapy, radiation
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Biological: anti-thymocyte globulin — Given IV
  Other Names: ATG; ATGAM; lymphocyte immune globulin; Thymoglobulin
Procedure: allogeneic bone marrow transplantation — Undergo allogeneic bone marrow transplant
  Other Names: bone marrow therapy, allogeneic; bone marrow therapy, allogenic; transplantation, allogeneic bone marrow; transplantation, allogenic bone marrow
Procedure: double-unit umbilical cord blood transplantation
Procedure: umbilical cord blood transplantation — Undergo allogeneic cord blood transplant
  Other Names: cord blood transplantation; transplantation, umbilical cord blood; UCB transplantation
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
Giving chemotherapy drugs, such as R115777, isotretinoin, cytarabine, and fludarabine, before a donor bone marrow transplant or an umbilical cord transplant helps stop the growth of cancer cells. It also helps stop the patient's immune system from rejecting the donor's stem cells. When the healthy stem cells from a donor are infused into the patient they may help the patient's bone marrow make stem cells, red blood cells, white blood cells, and platelets. This phase II trial is studying how well giving combination chemotherapy together with donor bone marrow or umbilical cord blood transplant works in treating children with newly diagnosed juvenile myelomonocytic leukemia

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the response rate of children with newly diagnosed juvenile myelomonocytic leukemia treated with R115777, isotretinoin, cytarabine, and fludarabine followed by allogeneic bone marrow or umbilical cord blood transplantation.

II. Determine the safety and toxicity of this regimen in these patients. III. Determine the tolerability of this regimen in these patients. IV. Determine the rate of 2-year event-free survival of patients treated with this regimen.

V. Determine whether prognostic subsets of these patients can be identified based on expression of clinical, genetic (NFI, monosomy 7, RAS gene), or hematopoietic characteristics.

OUTLINE: This is a multicenter study.

Patients may choose to receive upfront window induction therapy with oral R115777 twice daily on days 1-21. Treatment repeats every 28 days for 2 courses in the absence of disease progression or unacceptable toxicity.

Patients with progressive disease or stable disease with unacceptable hematopoietic recovery after 1 course proceed to induction chemotherapy. (R11577 portion of the study closed to accrual as of 08/2005)

All patients receive induction chemotherapy comprising oral isotretinoin once daily beginning on day 1 and fludarabine IV over 30 minutes and cytarabine IV over 4 hours on days 1-5. Treatment with fludarabine and cytarabine repeats every 28 days for 2 courses. Treatment with isotretinoin continues until allogeneic bone marrow or umbilical cord blood transplantation. Patients with progressive disease after 1 course proceed to transplantation.

After completion of isotretinoin, patients receive a preparative regimen comprising total body irradiation twice daily on days -7 to -4, cyclophosphamide IV over 2 hours on days -3 and -2, and anti-thymocyte globulin IV over 4-6 hours every 12 hours on days -3 to -1. Patients undergo allogeneic bone marrow or umbilical cord blood transplantation on day 0. Patients receive oral isotretinoin daily beginning on approximately day 60 and continuing for 1 year.

Patients are followed every 6 months for 5 years and then annually thereafter.

PROJECTED ACCRUAL: A maximum of 100 patients (18-46 receiving R115777 with induction chemotherapy [R11577 portion of the study closed to accrual as of 08/2005] and 27-54 receiving induction chemotherapy only) will be accrued for this study within 3.2 years.

ELIGIBILITY:
Inclusion Criteria:

* Newly diagnosed, previously untreated juvenile myelomonocytic leukemia
* Presenting with all of the following:

  * Absence of t(9;22) or bcr/abl by PCR
  * Absolute monocyte count greater than 1,000/mm^3
  * Less than 20% bone marrow blasts
* Presenting with at least 2 of the following:

  * Elevated F hemoglobin
  * Myeloid precursors in peripheral blood
  * WBC greater than 10,000/mm^3
  * Sargramostim (GM-CSF) hypersensitivity
* See Disease Characteristics
* Bilirubin no greater than 2.0 mg/dL
* ALT no greater than 3 times normal
* Creatinine no greater than 2 times normal
* No concurrent sargramostim (GM-CSF)
* No concurrent proton pump inhibitors

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Actual)
Dates: Start 2001-06; Primary Completion 2007-10 (Actual)

PRIMARY OUTCOMES:
Response rate (CR or PR) | Up to 6 years
  The response rates in the up-front window with respect to whether or not patients had vas activating mutations will also be estimated by proportions.
Duration of response | Up to 6 years
  Will be estimated by Kaplan-Meier method.
Progression-free survival | 2 years
  Will be estimated by Kaplan-Meier method.
Evaluation of prognostic importance of genetic marker | Up to 6 years
  Logrank test and Cox proportional hazards model will be applied.
Grade 3 or greater toxicities assessed using CTC version 2.0 | Up to 6 years

SECONDARY OUTCOMES:
Survival of patients receiving the window vs. not | Up to 6 years
Response status on end of course reports (pre vs.post) | Up to 6 years
  Signed-rank comparison of components of therapy will be done.

CONTACTS AND LOCATIONS:
Overall Officials: Robert Castleberry, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States

REFERENCES:
- [Derived] Stieglitz E, Gu CJ, Richardson M, Kita R, Santaguida MT, Ali KA, Strachan DC, Dhar A, Yam G, Anderson W, Anderson E, Hubner J, Tasian SK, Loh ML, Lacher MD. Tretinoin Enhances the Effects of Chemotherapy in Juvenile Myelomonocytic Leukemia Using an Ex Vivo Drug Sensitivity Assay. JCO Precis Oncol. 2023 Sep;7:e2300302. doi: 10.1200/PO.23.00302. PMID 37944074